CLINICAL TRIAL: NCT04468997
Title: Phase I Clinical Trial of Recombinant Anti-VEGF Human Monoclonal Antibody in the Treatment of Wet Age-related Macular Degeneration
Brief Title: The Study of Drug 601 in Patients With Wet Age-related Macular Degeneration (wAMD)
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 3SGJ601-AMD
Record Dates: First submitted 2020-07-08; First posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Wet Age-related Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- 601 dose level 1 treatment (Experimental)
  Interventions: Drug: Drug 601
- 601 dose level 2 treatment (Experimental)
  Interventions: Drug: Drug 601
- 601 dose level 3 treatment (Experimental)
  Interventions: Drug: Drug 601
- 601 dose level 4 treatment (Experimental)
  Interventions: Drug: Drug 601
- 601 dose level 5 treatment (Experimental)
  Interventions: Drug: Drug 601
- 601 dose level 6 treatment (Experimental)
  Interventions: Drug: Drug 601

INTERVENTIONS:
Drug: Drug 601 — Recombinant humanized anti-VEGF monoclonal antibody, drug 601(0.375mg), Vitreous injection, injection once;
  Arms: 601 dose level 1 treatment
Drug: Drug 601 — Recombinant humanized anti-VEGF monoclonal antibody, drug 601(0.75mg), Vitreous injection, injection once;
  Arms: 601 dose level 2 treatment
Drug: Drug 601 — Recombinant humanized anti-VEGF monoclonal antibody, drug 601(1.25mg), Vitreous injection, injection once;
  Arms: 601 dose level 3 treatment
Drug: Drug 601 — Recombinant humanized anti-VEGF monoclonal antibody, drug 601(2.5mg), Vitreous injection, injection once;
  Arms: 601 dose level 4 treatment
Drug: Drug 601 — Recombinant humanized anti-VEGF monoclonal antibody, drug 601(1.25mg), Vitreous injection, injection once every 4 weeks, three times continuously, then injection as needed within 9 months.
  Arms: 601 dose level 5 treatment
Drug: Drug 601 — Recombinant humanized anti-VEGF monoclonal antibody, drug 601(2.5mg), Vitreous injection, injection once every 4 weeks, three times continuously, then injection as needed within 9 months.
  Arms: 601 dose level 6 treatment

SUMMARY:
Multicenter study to evaluate the safety and tolerability in patients with wet Age-related macular degeneration (wAMD) treated with intravitreal recombinant humanized anti-VEGF monoclonal antibody

DETAILED DESCRIPTION:
According to the results of preclinical pharmacological research and clinical application of bevacizumab in ophthalmology Case, 601 will be developed as a drug candidate for the treatment of ocular diseases such as wAMD .Observe the safety and tolerability of the single and multiple doses of 601 in wAMD patients; study the pharmacokinetic characteristics of single and multiple doses of 601, Observe the Preliminary efficacy of 601 multiple injections with different doses in the treatment of patients with wAMD.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent form and willing to be visited at the time specified in the trial;
2. Age ≥45 years and age ≤ 80 years;
3. The study eye must meet the following criteria:

   * Diagnosis of wAMD;
   * The presence of an primary or recurrent active choroidal neovascular (CNV) lesions in subfovea and para-fovea secondary to AMD;
   * Total area of all types of lesions ≤30mm2 (12 optic disc areas)
   * Best EDTRS letter score between 19 and 78(Snellen equivalent of 20/400 to 20/32);
   * No optometric media opacity and pupil shrinkage.
4. Best EDTRS letter score ≥19 (Snellen equivalent of 20/400 or better) in the fellow eyes.

Exclusion Criteria:

Any of the following eye conditions:

1. Any eye has active ocular infections (e.g.,blepharitis, keratitis, scleritis, conjunctivitis);
2. History of vitreous hemorrhage in the study eye within 2 months before screening;
3. scarring, fibrosis, or atrophy below with fovea in the study eye;
4. Received any drug treatment for CNV within 120 days prior to screening;
5. History of any following surgery in the study eye (e.g. PDT, macular transposition, Glaucoma filtration, subfoveal photocoagulation, vitrectomy and transpupular hyperthermia, and other surgery at the submacular or others for AMD) within 3 months before screening;
6. CNV in the study eye associated with other ocular diseases such as pathologic myopia, eye trauma, etc
7. History or present of uncontrolled glaucoma, history of glaucoma filtering surgery in the study eye;
8. Subretinal hemorrhage in the study eye, and the bleeding area ≥ 50% area of the total lesion;
9. History of rhegmatogenous retinal detachment or macular hole retinal detachment (stage 3 or 4) , retinal detachment, retinal pigment epithelium tear or macular area traction and macular area preretinal membrane and PCV in the study eye;
10. The study eye has no lens( except intraocular lens) or posterior capsular rupture of the lens;

    Any of the following general condition are present:
11. Medicines with toxicity to the lens are being used or may be used during the study period;
12. History of allergy to fluorescein sodium and allergies to protein products for treatment or diagnosis, history of allergy to more than two drugs and/or non-drug factors, or suffering from allergic diseases now.
13. History of surgery within 1 months before screening; and/or unhealed wounds, ulcers or fractures currently;
14. Suffering from systemic infections and requiring oral, intramuscular or intravenous medication;
15. History of stroke, myocardial infarction within 6 months before screening;
16. Active diffuse intravascular coagulation and obvious bleeding tendency within 3 months before screening;
17. Systemic immune diseases;
18. Uncontrolled blood pressure control ;
19. Diabetic patients with uncontrolled blood sugar;
20. Any uncontrolled clinical problems (such as severe mental, neurological, cardiovascular, respiratory and other systemic diseases and malignant tumours);

    Any of the following laboratory tests abnormalities(23-25):
21. Renal function impairment (Cr is 1.5 times higher than the upper limit of normal values in the local laboratory) Liver dysfunction (ALT or AST is 2 times higher than the upper limit of normal value in the local laboratory).
22. Abnormal coagulation function (prothrombin time >= the upper limit of normal value for 3 seconds) and activated partial thromboplastin time >= the upper limit of normal value for 10 seconds);

    Patients with childbearing age with any of the following conditions:
23. Those who do not use effective contraceptive measures;

    The following are not excluded:
24. Pregnancy and lactation women (pregnancy is defined as urinary pregnancy test positive in this study);

    Any other conditions:
25. Participation in any other drug clinical trials (except vitamins and minerals) in the past 1 month before screening ;
26. Researchers think it needs to be ruled out.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Estimated)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
DLT | From Day 0 up to Day 14
  Incidence of dose-limiting toxicities up to the Day 14 visit
MTD | From Day 0 up to Day 56/112.
  Maximum tolerated dose

SECONDARY OUTCOMES:
Pharmacokinetic (PK) profile | From Day 0 up to 56/112 days
  Study the change of 601 drug concentration in the blood with time by mathematical principles and methods
Cmax | From Day 0 up to 56/112 days
  The maximum blood concentration after 601 drug enters the bloodstream
t1/2 | From Day 0 up to 56/112 days
  The half-life of drug 601, the time required for the terminal phase 601 drug concentration to drop by half
AUC | From Day 0 up to 56/112 days
  Area under the concentration-time curve, reflect the characteristics of the exposure of 601 drug in the body.
Vd | From Day 0 up to 56/112 days
  The proportional constant between the amount of 601 drug in the body and the blood concentration when the 601 drug achieves the dynamic balance in the body.
CL | From Day 0 up to 56/112 days
  Clearance rate of drug 601 from the central ventricle.
MRT | From Day 0 up to 56/112 days
  The average length of time that the 601 drug stays in the body.
λz | From Day 0 up to 56/112 days
  the ratio of the amount of elimination of 601 drug from the body per unit time to the total amount in the body
Biomarker | From Day 0 up to 56/112 days
  Detection of VEGF concentration.
Immunogenicity | From Day 0 up to 56/112 days
  Development of Anti-drug antibodies (ADA) after IVT injection of 601
CRT | From Day 0 up to 56/364 days
  Changes in central retina thickness (CRT) at all time points compared to the baseline
diseased region | From Day 0 up to 56/364 days
  Changes in the diseased region at all time points compared to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- BeiJing Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No